CLINICAL TRIAL: NCT00001387
Title: Phase I and Pharmacokinetic Trial of Paclitaxel (Taxol) Given as a 3-Hour Infusion in Pediatric Patients With Refractory Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940204; 94-C-0204
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Neoplasms
Keywords: Paclitaxel; Pediatric; Pharmacokinetics; Phase I; Toxicity
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
The objective of this trial is to determine the maximum tolerated dose and the toxicities of paclitaxel given as a short hour infusion in children with refractory malignancy.

DETAILED DESCRIPTION:
Paclitaxel is an active antitumor agent that has demonstrated a broad range of activity in preclinical and clinical studies. The optimal dose and schedule has not yet been determined in either adults or children. The objective of this trial is to determine the maximum tolerated dose and the toxicities of paclitaxel given as a short hour infusion in children with refractory malignancy. In addition, the pharmacokinetics of paclitaxel given in this way will be studied and both model-dependent and model-independent parameters will be determined.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed cancer (including leukemia) that is: Refractory to standard therapy (objective disease progression required) OR For which no standard therapy exists and patient is ineligible for potentially curative surgery.

PRIOR/CONCURRENT THERAPY:

Recovery from the toxic effects of prior therapy required.

Biologic Therapy: Not specified.

Chemotherapy: No prior taxanes. At least 3 weeks since myelosuppressive therapy (6 weeks since nitrosourea).

Endocrine Therapy: Not specified.

Radiotherapy: Prior extensive craniospinal or pelvic irradiation allowed.

Surgery: Ineligible for potential curative surgery.

Other: Prior bone marrow transplant allowed.

PATIENT CHARACTERISTICS:

Age: Over 1 to 21;

Performance status: ECOG 0-2;

Life expectancy: At least 8 weeks.

Hematopoietic: (except with leukemia, bone marrow involvement, history of bone marrow transplantation, or extensive prior radiotherapy).

Absolute granulocyte count at least 1,500/mm(3);

Platelet count at least 100,000/mm(3);

Hemoglobin at least 8.0 g/dL.

Hepatic:

Bilirubin no greater than 1.5 mg/dL;

AST less than 2 times normal.

Renal:

Creatinine no greater than 1.5 mg/dL OR;

Creatinine clearance at least 60 mL/min per square meter.

OTHER:

No concurrent anticonvulsant therapy.

No grade 2 or worse neuropathy.

No significant systemic illness (e.g., infection) that could compromise drug excretion or confuse assessment of toxicity.

Not pregnant or nursing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1994-09; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rowinsky EK, Donehower RC. The clinical pharmacology of paclitaxel (Taxol). Semin Oncol. 1993 Aug;20(4 Suppl 3):16-25. PMID 8102014
- [Background] Huizing MT, Keung AC, Rosing H, van der Kuij V, ten Bokkel Huinink WW, Mandjes IM, Dubbelman AC, Pinedo HM, Beijnen JH. Pharmacokinetics of paclitaxel and metabolites in a randomized comparative study in platinum-pretreated ovarian cancer patients. J Clin Oncol. 1993 Nov;11(11):2127-35. doi: 10.1200/JCO.1993.11.11.2127. PMID 7901342
- [Background] Kohn EC, Sarosy G, Bicher A, Link C, Christian M, Steinberg SM, Rothenberg M, Adamo DO, Davis P, Ognibene FP, et al. Dose-intense taxol: high response rate in patients with platinum-resistant recurrent ovarian cancer. J Natl Cancer Inst. 1994 Jan 5;86(1):18-24. doi: 10.1093/jnci/86.1.18. PMID 7505830